CLINICAL TRIAL: NCT01070771
Title: Does Routine Pressure Wire Assessment Influence Management Strategy at Coronary Angiography for Diagnosis of Chest Pain?
Acronym: RIPCORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Version 3 dated 01/10/2009; 5327 (Registry Identifier: UK Clinical Research Network Portfolio)
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2015-10

CONDITIONS: Coronary Artery Disease
Keywords: Pressure wire; Fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Radi pressure wire (pressure wire assessment) — Intracoronary insertion of pressure wire at the time of diagnostic angiography.
  Other Names: Radi pressure wire.

SUMMARY:
The use of coronary angiography to investigate patients at risk of coronary artery narrowings has become universal. In most cases, this investigation leads to a successful treatment plan with revascularisation recommended where appropriate. However in a substantial number of patients, the images taken of the coronary arteries can lead to diagnostic uncertainty. Increasingly, doctors are using devices called pressure wires to clarify the significance of coronary artery narrowings in order to tailor patient treatment on an individual basis.

The Radi pressure wire is well recognised as a reliable tool in assessing whether a narrowing is significant in functional terms, that is, does it significantly restrict blood flow to the heart muscle.It consists of a fine wire that is fed into individual major coronary arteries to measure pressure within the vessel itself. In conjunction with the images taken of the arteries, it is very useful in deciding how best to treat patients.

This study enrolls volunteers who are being investigated for stable cardiac-sounding chest pain and are undergoing a coronary angiogram. It will investigate whether the extra information gained from pressure wire assessment will change patients' treatment plan.

DETAILED DESCRIPTION:
The choice of management in an individual patient is determined largely by the presence and distribution of significant coronary narrowings. Usually, this significance is judged by the visual estimation of a narrowing on an angiogram. However, although this is the standard way of assessing coronary narrowings, it is now widely published that pressure wire measurements are more accurate because they assess the true physiological consequences of the narrowing. Interventional cardiologists now frequently use Fractional Flow Reserve (FFR) measurements to help them decide if arteries require stenting.The hypothesis for this study is that routine measurement of FFR in the main coronary arteries could provide diagnostic information above and beyond that obtained by an angiogram alone. This additional information may well then affect the choice of management in a proportion of these patients. For example, a narrowing considered to be significant angiographically may be shown to be insignificant with FFR, or vice versa.

Background

Coronary artery disease (CAD) is a major cause of morbidity and mortality in the United Kingdom. It accounts for approximately half of all cardiovascular related deaths annually and, according to statistics from the British Heart Foundation, CAD related expenditure was £3,500 million in 2003 alone. Much effort has been placed on improving methods that detect and assess the severity of CAD and facilitate more rapid and appropriate management for CAD patients. Once diagnosed, CAD may be treated in 3 ways: (1)tablets alone, (2)tablets plus angioplasty with stents or (3) tablets plus coronary artery bypass graft surgery (CABG). The method of choice depends primarily on the extent and severity of disease at the time of coronary angiography. Coronary angiography is the current conventional method for the diagnosis of CAD and is used in the assessment of disease severity. For the angiographic procedure,vascular access is secured via the femoral artery or radial artery route and a dye is injected into the coronary artery blood vessels. The progress of the dye through the coronary blood vessels provides a visual assessment of where narrowings are present in the coronary arteries.

Where there is thought to be significant flow obstruction, particularly in symptomatic patients, one of the above three treatments will be offered.

While coronary angiography has revolutionised the management of CAD, the procedure is not without limitation. The purely visual assessment of disease severity with coronary angiography is subjective and patient management can depend on the cardiologist reviewing the films. Many such narrowings can be graded 'moderate' severity and deciding whether these are of haemodynamic significance is notoriously difficult by angiography alone. In recent years, the Radi pressure wire has been shown to provide accurate physiological haemodynamic data about coronary narrowings. Furthermore, the FFR measurement derived predicts clinical outcome, hence giving a 'cut-off' measurement for severity of disease that correlates with the requirement for revascularisation with either stents or surgery. Thus FFR is now frequently used in clinical practice by interventional cardiologists to decide if narrowings require treatment. However, the majority of diagnostic angiography in the UK is performed by non-interventional cardiologists who do not currently have access to the pressure wire technology. In this study, we speculate that if we measure the FFR routinely in all the main coronary arteries of patients undergoing coronary angiography the FFR data obtained may affect the angiogram-derived management of some patients in terms of the choice of tablets/stents/CABG. For example, some narrowings that look significant angiographically may not be haemodynamically important by FFR and vice versa. Clearly this could make a difference between revascularising a patient or not.

Research Aims

To evaluate:

1. The degree of correlation between standard angiographic assessment of the coronary arteries and pressure wire assessment of the main arteries.
2. To determine whether the FFR data would influence the management strategy for patients as derived only on the basis of the angiogram (which represents clinical practice).

Methods and Design

The study will recruit 200 patients listed for diagnostic coronary angiography performed by a non-interventional cardiologist.

Methodology 1: In Catheter Laboratory

* All patients will receive an information sheet after initial invitation to take part.
* Written informed consent will be obtained.
* Patients will undergo coronary angiography in a routine manner.
* The non-interventional cardiologist in charge of the patient's care will analyse the pictures and grade the outcome in the manner shown in table 1. He/she will formulate a management plan consistent with their routine clinical practice and independent of subsequent pressure wire data. This management plan will be documented in the CRF. He/she will then take no further part in the procedure.

Table 1

1. Are there significant stenoses (>70% by eyeball) in the major epicardial vessels (i.e. main coronaries or any branch of >2.25mm)
2. Recommend revascularisation or medical/conservative treatment
3. If revascularisation: recommended strategy for referral (Percutaneous Coronary Intervention (PCI) or CABG?) and which vessels (i.e. LAD + RCA etc) represent targets for that revascularisation

   * The management strategy will be recorded according to the following options:

     1. medical;
     2. PCI
     3. CABG
   * Data will also be collected in regard to vessels as targets (i.e. which vessels require stent/graft)
   * If the non-interventional cardiologist cannot make a plan they can allocate the patient to a fourth category in which "more data are required". Such patients are generally then referred for further non-invasive stress imaging or even for a pressure wire.
   * FFR measurements will then be undertaken by a consultant interventional cardiologist
   * Additional screening time and contrast use accrued during FFR measurements will be recorded.
   * The patient will be given 70units/kg heparin i.a. or i.v. prior to passage of the pressure wire
   * A pressure wire will be introduced into the distal third of all patent major epicardial coronary arteries and branches of >2.25mm with TIMI 3 flow.
   * FFR measurements will be taken using either intracoronary or intravenous adenosine according to local conventional practice and operator preference.
   * The protocol mandates i.v. adenosine for ostial LM stem and ostial RCA stenoses.
   * Where i.c. adenosine bolus is employed, the minimum data required by the study is: 1 baseline FFR without adenosine and 2 boluses with at least 50mcg adenosine.
   * An angiogram will be acquired before the first adenosine measurement to document satisfactory engagement of the guiding catheter and the position of the measurement in each vessel
   * The minimum FFR reading will be taken in each case
   * FFR readings of <0.8 will be considered as representing haemodynamic significance as per FAME protocol
   * Once the FFR data are derived the procedure will be finished and haemostasis will be achieved in the normal manner
   * Provided the angiogram-derived management plan has been recorded in the CRF then the FFR data can then be revealed to the non-interventional cardiologist. The management plan will then be recorded in the light of the FFR data using the same categories and dataset as previously.
   * The non-interventionalists will then manage the patient as they see fit

Analysis

PRIMARY ENDPOINT Estimation of number of cases where FFR data results in a change in the management strategy the revascularisation strategy (number of vessel requiring treatment and/or PCI vs medical vs CABG)

Potential Clinical Value

If this study proves its hypothesis, it will suggest that coronary angiography would be better supported by routine pressure wire assessment in order to tailor revascularisation strategies for individual patients more accurately. The result of this study will carry important clinical implications if the study hypothesis is proven.... not least in terms of potential patient benefit. The current widely held practice of diagnostic test followed by either (i) referral for revascularisation or, (ii) in the case of equivocal angiographic results, referral for stress imaging to look for objective evidence of ischaemia followed by referral for revascularisation where positive could be rendered obsolete by diagnostic angiography performed by interventional cardiologists with FFR availability and the ability to perform PCI at the same sitting where appropriate.

The study may generate the hypothesis that such routine FFR measurement will not only be of benefit to patients but also be cost-effective if there would have been fewer interventions overall (ie less CABG + PCI) or fewer expensive interventions (i.e. less CABG versus PCI)?

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for elective coronary angiography under a non-interventional cardiologist for the investigation of chest pain thought to be of cardiac origin.
* There is no requirement for a test demonstrating objective evidence of myocardial ischaemia because this study aims to recruit consecutive patients in real world current practice
* Written informed consent
* No participation in other studies

Exclusion Criteria:

* Previous coronary artery bypass graft surgery
* Acute coronary syndrome at presentation
* Diagnostic angiography or percutaneous coronary intervention within the previous 12 months
* Contraindication to adenosine
* Severe valve disease
* Creatinine >180
* Life threatening comorbidity
* Diagnostic angiogram showing "normal" coronary arteries defined as no coronary stenosis of >30% by visual estimate in any epicardial vessel of >2.25mm diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2008-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Curzen, BM(Hons) PhD FRCP, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (10):
- Dr Colm Hanratty, Belfast, Ireland
- United Kingdom (9):
  - Dr Alex Hobson, Portsmouth, Hampshire
  - Dr Dan McKenzie, Taunton, Somerset
  - Royal Sussex County Hospital, Brighton
  - Dr Kamal Chitkara, Derby
  - West of Scotland Regional Heart & Lung Centre, Glasgow
  - Dr Steve Wheatcroft, Leeds
  - Freeman Hospital, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford
  - Southampton General Hospital, Southampton

REFERENCES:
- [Result] Curzen N, Rana O, Nicholas Z, Golledge P, Zaman A, Oldroyd K, Hanratty C, Banning A, Wheatcroft S, Hobson A, Chitkara K, Hildick-Smith D, McKenzie D, Calver A, Dimitrov BD, Corbett S. Does routine pressure wire assessment influence management strategy at coronary angiography for diagnosis of chest pain?: the RIPCORD study. Circ Cardiovasc Interv. 2014 Apr;7(2):248-55. doi: 10.1161/CIRCINTERVENTIONS.113.000978. Epub 2014 Mar 18. PMID 24642999
- [Derived] Bashar HAB, Saunders A, Alaour B, Gerontitis D, Hinton J, Karamanou D, Kechagioglou G, Olsen S, Onwordi E, Pope M, Zingale A, Nicholas Z, Golledge P, Escaned J, Ali Z, Curzen N. Systematic coronary physiology improves level of agreement in diagnostic coronary angiography. Open Heart. 2023 May;10(1):e002258. doi: 10.1136/openhrt-2023-002258. PMID 37130658
- [Derived] Stables RH, Mullen LJ, Elguindy M, Nicholas Z, Aboul-Enien YH, Kemp I, O'Kane P, Hobson A, Johnson TW, Khan SQ, Wheatcroft SB, Garg S, Zaman AG, Mamas MA, Nolan J, Jadhav S, Berry C, Watkins S, Hildick-Smith D, Gunn J, Conway D, Hoye A, Fazal IA, Hanratty CG, De Bruyne B, Curzen N. Routine Pressure Wire Assessment Versus Conventional Angiography in the Management of Patients With Coronary Artery Disease: The RIPCORD 2 Trial. Circulation. 2022 Aug 30;146(9):687-698. doi: 10.1161/CIRCULATIONAHA.121.057793. Epub 2022 Aug 10. PMID 35946404

RESULTS

PARTICIPANT FLOW:
Groups:
- Radi Pressure Wire: Assessment of physiological significance of coronary artery narrowings by measurement of blood flow limitation across lesion.
Period: Overall Study
Arm/Group | Radi Pressure Wire
Started | 203 (September 2008)
Completed | 200 (August 2012)
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radi Pressure Wire
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 149
Region of Enrollment [Number; unit: participants]
  United Kingdom | 200

OUTCOME MEASURES:

1. Primary Outcome: Estimation of Number of Cases Where FFR Data Results in a Change in the Management Strategy (Number of Vessel Requiring Treatment and/or PCI vs Medical vs CABG)
Description: This outcome measure was assessing agreement in the management plan (MP) derived from angiographic assessment alone compared to a MP derived from angiographic assessment plus the use of FFR data acquired at the time of angiography. The study assessed the proportion of cases in which the angiogram directed MP changed after FFR data were disclosed.
Time Frame: Up until hospital discharge. Most cases were day cases but no specific data relating to length of stay collected.
Measure: Number; unit: participants
Arm/Group | Radi Pressure Wire
Number analyzed (Participants) | 200
participants
  Agreement with management plan | 147
  Change in management plan after FFR | 53
  Recommended medical treatment alone | 72
  Revascularisation was advised after FFR | 9
  Optimal medical therapy recommended after FFR | 89
  Recommended revascularisation after angiogram | 25
  Recommendation of PCI after angio assessment | 90
  Of the 90 FFR detected no significant stenosis | 24

2. Secondary Outcome: To Determine the Level of Agreement in Management Plans Regarding the Significance of Coronary Artery Narrowings When Comparing the MP Acquired by Standard Angiographic Assessment Alone and a MP Acquired Using Angiographic Assessment Plus FFR Data.
Description: This compared the number of vessels in which there was a discrepant result in relation to angiographically and FFR defined significance. Angiographic significance was visually assessed by operators whereas the pressure wire provided objective data as to a narrowing's significance: an FFR reading of <0.8 indicated a significant restriction in blood flow with a recommendation for revascularisation.
  The difference in indication for revascularisation of each major coronary artery was also judged according to angiogram alone compared with angiogram plus FFR dtaa.
Time Frame: Up to hospital discharge. Most were day case procedures but no specific data relating to discharge was collected.
Measure: Number; unit: participants
Arm/Group | RADI Pressure Wire
Number analyzed (Participants) | 200
participants
  Number of vessels significantly changed after FFR | 64
  No significant CAD after angiography alone | 81
  Of the 81, significant FFR (<0.8) | 18
  No haemodynamically signifiacnt CAD after FFR | 89
  Of the 89, angio labelled as single vessel disease | 24
  of the 89, angio labelled as 2 vessel disease | 1
  of the 89, angio labelled as 3 vessel disease | 1
  significant 3 vessel disease at angio:negative FFR | 1

ADVERSE EVENTS:
Description: Only serious adverse events were collected
Arm/Group | RADI Pressure Wire
Serious Adverse Events (participants affected / at risk) | 3/200
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RADI Pressure Wire (N=200)
Vessel occlusion (Cardiac disorders) | 1 (1) — In one patient, the operator crossed a tightly stenosed right coronary artery with the pressure wire but this vessel subsequently occluded, leading to emergency PCI and a troponin rise to 5.88mcg/L.
Coronary artery dissection (Cardiac disorders) | 1 (1) — a second case, the pressure wire manipulation in the left anterior descending artery led to coronary artery dissection and the patient underwent emergency CABG surgery, which was subsequently complicated by a deep vein thrombosis.
Ventricular fibrillation (Cardiac disorders) | 1 (1) — In one patient there was an episode of ventricular fibrillation during FFR assessment of the RCA and the operator decided not to proceed to further measurements .
Deep vein thrombosis (Vascular disorders) | 1 (1) — Patient underwent emergency CABG and subsequently went on to experience DVT

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days